CLINICAL TRIAL: NCT04382872
Title: Investigation of Follicular Fluid Exosome miRNA in Young and Aged Women During Oocyte Maturation
Brief Title: Follicular Fluid Exosome miRNA During Oocyte Maturation
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2019.137
Record Dates: First submitted 2020-04-23; First posted 2020-05-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Oocyte Maturation
Keywords: oocyte maturation; in vitro maturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Folliculogenesis involves the recruitment of primordial follicles into a group of growing follicles in which eventually one follicle is selected, matured and ovulated. Complex endocrine and intra-ovarian paracrine interactions occur to create a changing intra-follicular hormonal milieu suitable for oocyte development. However, this oocyte developmental competence and to undergo fertilization and embryogenesis is impaired in aged women. Diminished ovarian function is generally attributed to decreased quantity and quality of oocytes and their surrounding granulosa cells during ovarian aging, although the underlying mechanisms remain unclear.

The aim of the study is to investigate the miRNA in (follicular fluid) FF exosome in young and aged women and their relationship to egg maturation.

DETAILED DESCRIPTION:
In recent decades, demographic and socioeconomic factors have resulted in marked changes in human society that include postponement of child bearing and a subsequent rise in mean age at first childbirth. Aged women have more reproductive problems (including menstrual irregulation and decreased ovarian reserve as reflected by reduced anti-mullerian hormone (AMH)) and their oocytes are often of lower quality when compared to younger women.

Folliculogenesis involves the recruitment of primordial follicles into a group of growing follicles in which eventually one follicle is selected, matured and ovulated. Complex endocrine and intra-ovarian paracrine interactions occur to create a changing intra-follicular hormonal milieu suitable for oocyte development. However, this oocyte developmental competence, defined as the ability of the oocyte to complete follicular development, and to undergo fertilization and embryogenesis is impaired in aged women. Age-related decline in female fertility is mainly driven by ovarian aging, or diminished ovarian function associated with age. Diminished ovarian function is generally attributed to decreased quantity and quality of oocytes and their surrounding granulosa cells during ovarian aging, although the underlying mechanisms remain unclear. Transcription studies have suggested indirectly that some age-related changes in oocyte gene expression and cell to cell communication may involve epigenetic machinery.

Ovarian follicle may be one of the best models in human for exosome study considering the role of the granulosa cells and follicular fluid for oocyte maturation. In the ovarian follicle, follicular fluid (FF) exosome may play an important mediated communication role between the oocyte and surrounding granulosa cells.

The aim of the study is to investigate the miRNA in (follicular fluid) FF exosome in young and aged women and their relationship to egg maturation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20 to 45;
2. BMI > 19 & < 35;
3. Women who is planning to perform invitro fertilization (IVF) together with intracytoplasmic sperm injection (ICSI) for their fertility problems

Exclusion Criteria:

1. Positive pregnancy test before taking study medications;
2. Women with BMI>35 kg/m2;
3. Women with known chromosomal translocation, recurrent abortions or those carrying Fragile X;
4. Women with endometriosis

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — this study required the subject to provide follicular fluid and immature oocyte, and therefore the subjects must be female
Study Population: women undergoing oocyte retrieval treatment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
RNA-sequencing | through study completion, an average of 2 years
  1) To identify for the first time FF exosome miRNAs in mature and immature follicles in young and aged women by RNA-sequencing (RNA-seq).
quantitative real-time polymerase chain reaction | through study completion, an average of 2 years
  2) To verify the identified FF exosome miRNAs in mature and immature follicles in young and aged women and investigate their expression in the corresponding granulosa cells by quantitative real-time polymerase chain reaction (qRT-PCR).

SECONDARY OUTCOMES:
fertilization and pregnancy rate | through study completion, an average of 2 years
  3) To observe the effect of the identified specific FF exosome miRNAs on oocyte maturation (by IVM) and assess the association of the miRNAs on fertilization and pregnancy rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong